CLINICAL TRIAL: NCT00887367
Title: A Study to Investigate Potential Interactions Between GSK598809 and Ethanol in Healthy Subjects
Brief Title: EtOH Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 106591
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Substance Dependence
Keywords: Healthy volunteers; Substance dependence; Alcohol dependence
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism | interventions — GSK598809; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo to match GSK598809 (Placebo Comparator): Placebo to match GSK598809.
  Interventions: Drug: GSK598809
- Placebo to match ethanol infusion (Placebo Comparator): Glucose solution to be given in the same way as ethanol.
  Interventions: Other: Ethanol

INTERVENTIONS:
Drug: GSK598809 — Two 175 mg doses of GSK598809 will be given.
  Arms: Placebo to match GSK598809
Other: Ethanol — A constant ethanol level of 0.6 g·L-1 for five hours will be given to the subjects intravenously. This level shows significant CNS effects, without causing too many inadvertent events. Furthermore this level is considered safe as it is just above the legal driving limit in the Netherlands (i.e. 0.5 g·L-1) and these levels are routinely achieved during social drinking. Moreover, this level leaves enough room for CNS-impairment without compromising safety, in case of a (supra-) addictive drug-alcohol interaction.
  Arms: Placebo to match ethanol infusion

SUMMARY:
This study will investigate the possible effects of alcohol in combination with GSK598809 on the central nervous system in 20 healthy male and female volunteers, between 18 and 65 years of age.

During 4 separate study periods subjects will receive the following treatment combinations: Alcohol + GSK598809, alcohol + placebo drug, placebo infusion + GSK598809, and placebo infusion + placebo drug. A placebo is a pill or liquid infusion which contains no drug or alcohol; it is a dummy version. Therefore it is administered in the same way that either the study drug or ethanol is depending on which placebo it is. All study drugs are administered in a random order and both the doctor and the participant are not aware of the treatment combination. However treatment combinations will be available at the end of the study or in case of an emergency. GSK598809 is administered orally and alcohol is administered per infusion. The duration of the infusion is 5 hours, during which approximately 75 grams of alcohol is infused, which is comparable to less than one bottle of wine.

DETAILED DESCRIPTION:
This is a blinded, randomised, placebo-controlled, double-dummy, four-period crossover study to investigate the psychomotor and cognitive effects of GSK598809 alone and in combination with ethanol in healthy subjects.

A sufficient number of subjects, approximately 20 healthy (18 to 65 years) male and female subjects will be enrolled. Occasional smokers who are non-daily smokers may be enrolled in the study, but will not be permitted to smoke whilst in the unit.

Subjects will be screened by medical history, physical examination and routine laboratory tests within three weeks before the start of the study. Within three weeks or on Day -1 they will have a training session to get familiar with the pharmacodynamic tests.

There will be four crossover sessions. All study occasions/sessions will be performed in the same way. The duration of each treatment session is 5 study days. Subjects will report to the clinic during the evening of Day -1 in a fasted condition and will remain in the clinic for two overnight stays. A short study introduction will be given followed by admission procedures. Dinner will be served after the collection of blood samples for laboratory safety tests.

On morning of study day 1, approximately 08:00hrs two intravenous cannulae (one cannula for blood sampling and another cannula for infusion of the ethanol/placebo) will be inserted. Before the start of the infusion a light breakfast will be given. The alcohol infusion will start in the morning, between approximately 09:30hr and 10:00hr and will take place for five hours, followed by a three-hour infusion-free washout period. GSK598809 or matching placebo will be administered orally 30 minutes after the start of the alcohol infusion. A standardised lunch will be given at approximately 3.5 hours post dose and dinner approximately 9 hours post dose.

Subjects will be discharged after the completion of study assessments and AE review on Day 2 and if deemed appropriate by the investigator or designee. Study Days: 3 and 4 will be outpatient visits for collection of pharmacokinetic samples and AE review.

During each session, a range of central nervous system (CNS) functions will be tested frequently, using a validated CNS-battery, CHDR Neurocart. In addition, pharmacokinetic measurements will be taken for plasma levels of GSK598809 and GSK685249 (GSK598809 metabolite). Pharmacokinetic measures will also be taken for breath alcohol and blood alcohol levels.

There will be a washout period of at least five days between treatment sessions. The follow up visit will take place approximately 7 days post final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy.
* Occasional non-daily smokers.
* Willing to use appropriate contraception method.
* Weight more than 50 kg.
* BMI within the range 18 - 30 kg/m2.

Exclusion Criteria:

* Pregnant or breast feeding female.
* Daily smoker.
* Asthma or a history of asthma.
* Abuse of drugs or alcohol.
* Psychiatric illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09-29 (Actual); Primary Completion 2008-12-03 (Actual); Study Completion 2008-12-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Vital sign measurement, 12 lead ECG and telemetry, safety laboratory sampling including prolactin and lipid measurements, Barnes Akathesia Scale (BAS), Simpson-Angus Scale (SAS) and Abnormal Involuntary Movement Scale (AIMS). | Screening: BAS, SAS and AIMS (as training only), 12 lead ECG, vital signs and clinical labs. All will be measured throughout dosing day (Day 1), day 2, 3: vital signs, day 4: vital signs, clinical labs, follow up: clinical labs, vital signs, 12 lead ECG
Pharmacokinetics: breath ethanol concentrations, blood ethanol concentrations, main pharmacokinetic parameters of GSK598809 and its metabolite (GSK685249) AUC∞, Cmax, Tmax and t½. | All will be measured throughout day 1, PK blood sampling for GSK598809 and GSK685249 will also be collected on Day 2, 3 and 4.
Pharmacodynamic: saccadic eye movements, smooth pursuit eye movements, body sway, adaptive tracking, Visual Verbal Learning Test (VVLT). | Saccadic eye movement, smooth pursuit eye movements, body sway and adaptive tracking measured at set intervals between 1.5hrs pre dose to 7.5hrs post dose. VVLT administered between 0.5hrs post dose to 3.5hrs post dose.

SECONDARY OUTCOMES:
Pharmacodynamic/biomarker endpoints: saccadic eye movements, visual analogue scales (VAS B&L) according to Bond & Lader, Visual Analogue Scales for 'alcohol effects' (VAS 'Alcohol Effects'). | Saccadic eye movements at time points as given above. VAS B&L and VAS 'Alcohol Effects' at following time points: -1.5, 0.5, 1.5, 2.5, 3.5, 4.5, 5.5, 6.5, 7.5 hrs post dose.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Leiden, Netherlands

REFERENCES:
- [Background] te Beek ET, Zoethout RW, Bani MS, Andorn A, Iavarone L, Klaassen ES, Fina P, van Gerven JM. Pharmacokinetics and central nervous system effects of the novel dopamine D3 receptor antagonist GSK598809 and intravenous alcohol infusion at pseudo-steady state. J Psychopharmacol. 2012 Feb;26(2):303-14. doi: 10.1177/0269881111431750. Epub 2012 Jan 4. PMID 22219221
- See also: Results for study 106591 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/106591?search=study&search_terms=106591#rs